CLINICAL TRIAL: NCT05987397
Title: Clinical Multi-center Study of Mitochondrial Brain Protective Agent Idebenone in the Prevention of Post-stroke Epilepsy
Brief Title: Exploring the Preventive Effect of Mitochondrial Protective Agent Idebenone on Post-stroke Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Feng, MD, PhD, Associate Professor Vice Director of Neurology Teaching and Research Office, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202306124
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Post Stroke Epilepsy
Keywords: post-stroke epilepsy; idebenone
MeSH Terms: interventions — idebenone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Idebenone short-term treatment group (Experimental): The patient received oral idebenone 30 mg three times a day after stroke for a total course of 14 days (acute phase).
  Interventions: Drug: idebenone 30 mg for 14 days
- Group B: Idebenone long-term treatment group (Experimental): The patient will be treated with oral idebenone 30 mg three times a day after stroke for a total course of 3 months.
  Interventions: Drug: idebenone 30 mg for 3 months

INTERVENTIONS:
Drug: idebenone 30 mg for 14 days — The patient received oral idebenone 30 mg three times a day after stroke for a total course of 14 days (acute phase).
  Arms: Group A: Idebenone short-term treatment group
Drug: idebenone 30 mg for 3 months — The patient will be treated with oral idebenone 30 mg three times a day after stroke for a total course of 3 months.
  Arms: Group B: Idebenone long-term treatment group

SUMMARY:
According to the random number table, all patients were divided into short-term treatment group, long-term treatment group and non-intervention stroke control group according to the proportion of (1:1:1) epilepsy disease modifier idebenone. Patients in the short-term treatment group will take idebenone for a total course of 14 days (acute period) after stroke, and patients in the long-term treatment group will take idebenone for a total course of 3 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital within 24 hours of stroke symptoms and diagnosed with stroke (including cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, intracranial venous sinus thrombosis, etc.) after relevant examinations;
* Able to cooperate with the inspection;
* Sign the informed consent form.

Exclusion Criteria:

* History of epilepsy before stroke;
* A history of serious comorbidities that may lead to seizures (including malignant tumors, specific autoimmune diseases, severe electrolyte abnormalities, end-stage renal disease, and severe head trauma);
* Secondary stroke caused by head trauma or surgery;
* Other patients that the researchers think need to be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with epilepsy after stroke | At the time of enrollment
  Count the number of people with post-stroke epilepsy
The proportion of patients with epilepsy after stroke | 24 weeks after enrollment
  Count the number of people with post-stroke epilepsy
The proportion of patients with epilepsy after stroke | 48 weeks after enrollment
  Count the number of people with post-stroke epilepsy

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | At the time of enrollment
  The minimum value is 0, the maximum value is 24, the higher score indicates the more severe neurological impairment in stroke patients
National Institutes of Health Stroke Scale (NIHSS) | 24 weeks after enrollment
  The minimum value is 0, the maximum value is 24, the higher score indicates the more severe neurological impairment in stroke patients
National Institutes of Health Stroke Scale (NIHSS) | 48 weeks after enrollment
  The minimum value is 0, the maximum value is 24, the higher score indicates the more severe neurological impairment in stroke patients
Hamilton Anxiety Scale (HAMA) | At the time of enrollment
  The minimum value is 0, the maximum value is 56, the higher score indicates a great likelihood of anxiety
Hamilton Anxiety Scale (HAMA) | 24 weeks after enrollment
  The minimum value is 0, the maximum value is 56, the higher score indicates a great likelihood of anxiety
Hamilton Anxiety Scale (HAMA) | 48 weeks after enrollment
  The minimum value is 0, the maximum value is 56, the higher score indicates a great likelihood of anxiety
Hamilton Depression Scale (HAMD) | At the time of enrollment
  The minimum value is 0, the maximum value is 77, the higher score indicates a great likelihood of depression
Hamilton Depression Scale (HAMD) | 24 weeks after enrollment
  The minimum value is 0, the maximum value is 77, the higher score indicates a great likelihood of depression
Hamilton Depression Scale (HAMD) | 48 weeks after enrollment
  The minimum value is 0, the maximum value is 77, the higher score indicates a great likelihood of depression
Pittsburgh sleep quality index (PSQI) | At the time of enrollment
  The minimum value is 0, the maximum value is 21, the higher score indicates poorer sleep quality
Pittsburgh sleep quality index (PSQI) | 24 weeks after enrollment
  The minimum value is 0, the maximum value is 21, the higher score indicates poorer sleep quality
Pittsburgh sleep quality index (PSQI) | 48 weeks after enrollment
  The minimum value is 0, the maximum value is 21, the higher score indicates poorer sleep quality
Stroke specific quality of life scale (SS-QOL) | At the time of enrollment
  The minimum value is 38, the maximum value is 190, the higher score indicates better quality of life
Stroke specific quality of life scale (SS-QOL) | 24 weeks after enrollment
  The minimum value is 38, the maximum value is 190, the higher score indicates better quality of life
Stroke specific quality of life scale (SS-QOL) | 48 weeks after enrollment
  The minimum value is 38, the maximum value is 190, the higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China